CLINICAL TRIAL: NCT02678689
Title: A Phase 2, Open-Label, Multicenter Study to Evaluate Safety, Tolerability, and Efficacy of Intracerebroventricular BMN 190 in Pediatric Patients < 18 Years of Age With CLN2 Disease
Brief Title: A Safety, Tolerability, and Efficacy Study of BMN 190 in Pediatric Patients < 18 Years of Age With CLN2 Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190-203
Record Dates: First submitted 2016-01-15; First posted 2016-02-10 (Estimated); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-11

CONDITIONS: Jansky-Bielschowsky Disease; Batten Disease; Late-Infantile Neuronal Ceroid Lipofuscinosis Type 2; CLN2 Disease; CLN2 Disorder
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses | interventions — cerliponase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- BMN 190 recombinant human tripeptidyl peptidase-1 (rhTPP1) (Experimental): An age-appropriate dose of BMN 190 administered via intracerebroventricular (ICV) infusion every other week (qow) for a duration of 144 weeks.
  Interventions: Biological: BMN 190 recombinant human tripeptidyl peptidase-1 (rhTPP1); Device: Intracerebroventricular access device

INTERVENTIONS:
Biological: BMN 190 recombinant human tripeptidyl peptidase-1 (rhTPP1)
  Other Names: recombinant human tripeptidyl peptidase-1 (rhTPP1); cerliponase alfa; Brineura®
Device: Intracerebroventricular access device — Surgical implantation of an MRI compatible ICV access device in the lateral ventricle of the right hemisphere is required for administration of study drug.

SUMMARY:
This Phase 2 open-label, multicenter study will evaluate the safety, tolerability, and efficacy of BMN 190 intracerebroventricular (ICV) administration every other week (qow) for a period of 144 weeks, in patients with CLN2. The study is designed to assess disease progression in CLN2 patients treated with BMN 190 compared to natural history data from untreated historical controls.

DETAILED DESCRIPTION:
BMN 190 is a recombinant form of human tripeptidyl peptidase 1 (TPP1), the enzyme deficient in patients with CLN2 diseases (also known as classical late-infantile CLN2, cLINCL, or Jansky-Bielschowsky disease), a form of Batten Disease. As an enzyme replacement therapy (ERT), BMN 190 is designed to help restore TPP1 enzyme activity. BMN 190 is designed to reduce the progressive, pathologic accumulation of lysosomal storage material. 190-203 is a Phase 2 open-label, multicenter study that will evaluate the safety, tolerability, and efficacy of BMN 190 in pediatric patients < 18 years of age with CLN2 disease. Study drug dosing will be determined by the patient's age and administered via intracerebroventricular (ICV) infusion every other week (qow), for a duration of 144 weeks.

ELIGIBILITY:
Enrollment is complete.

Inclusion Criteria:

* Diagnosis of CLN2 disease as determined by TPP1 enzyme activity (dried blood spot) in the fibroblasts and leukocytes available at Screening
* Quantitative clinical assessment of the Hamburg motor-language aggregate score 3-6 at Screening on CLN2 disease motor-language scale, as defined in the Ratings Assessment Guideline
* < 18 years of age at the time of informed consent
* Written informed consent from parent or legal guardian and assent form subject, if appropriate
* Males and females who are of reproductive age should practice true abstinence, defined as no sexual activity, during the study and for 6 months after the study has been completed (or withdrawal from the study). If sexually active and not practicing true abstinence, males and females of reproductive age must use a highly effective method of contraception while participating in the study.
* Ability to comply with protocol required assessments (ICV implantation, drug administration, laboratory sample collection, electroencephalogram (EEG), electrocardiogram (ECG),magnetic resonance imaging (MRI), etc.)

Exclusion Criteria:

* Presence of another inherited neurological disease, e.g., other forms of CLN or seizures unrelated to CLN2 disease (patients with febrile seizures may be eligible)
* Presence of another neurological illness that may have caused cognitive decline (e.g., trauma, meningitis, hemorrhage) or interference with disease rating (autism) before Screening
* Presence of percutaneous feeding tube placement prior to enrollment
* Has received stem cell, gene therapy, or ERT
* Presence of contraindications for neurosurgery (e.g., congenital heart disease, severe respiratory impairment, or clotting abnormalities)
* Presence of contraindications for MRI scans (e.g., cardiac pacemaker, metal fragment or chip in the eye, aneurysm clip in the brain)
* Episode of generalized motor status epilepticus within 4 weeks before the First Dose visit
* Severe infection (e.g., pneumonia, pyelonephritis, or meningitis) within 4 weeks before the First Dose visit (enrollment may be postponed)
* Presence of ventricular abnormality (hydrocephalus, malformation)
* Presence of ventricular shunt
* Has known hypersensitivity to any of the components of BMN 190
* Has received any investigational mediation within 30 days before the first infusion of study drug or is scheduled to receive any investigational drug other than BMN 190 during the course of the study
* Has a medical condition or extenuating circumstance that, in the opinion of the investigator, might compromise the subject's ability to comply with the protocol required testing or procedures or compromise the subject's well being, safety, or clinical interpretability
* Pregnancy any time during the study; a female subject judged by the investigator to be of childbearing potential will be tested for pregnancy

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2016-01-22 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (4):
- Nationwide Children's Hospital, Columbus, Ohio, United States
- Universitaetsklinikum Hamburg-Eppendorf, Hamburg, Germany
- Children's Hospital Bambino Gesù,IRCCS, Rome, Piazza, Italy
- Great Ormond Street Childrens Hospital, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study 190-203 was conducted at 4 clinic sites:One each in Germany, Italy, the United Kingdom and the United States.
  The comparator group for determination of the primary efficacy outcome measures in this study was comprised of 29 Natural History (NH) subjects with late-infantile neuronal ceroid lipofuscinosis disease, also known as classical late-infantile CLN2, cLINCL, or Jansky-Bielschowsky disease, a form of Batten Disease (CLN2) disease selected from the DEM-CHILD database (NCT04613089).
Pre-assignment Details: A total of 14 participants were enrolled and treated in study 190-203. 13 participants completed the study, and 1 participant withdrew to receive treatment commercially.
  The 190-203 study required enrollment of at least 10 participants, including at least 5 participants with a combined ML score >= 5 points (mild or pre-symptomatic disease), at least 5 participants with a ML score < 5points (moderate disease), and at least 5 participants < 2 years of age.
Groups:
- BMN 190-203: BMN 190 was administered by continuous Intracerebroventricular (ICV) infusion at the rate of 2.5 mL/hour for approximately 4 hours every 14 (+/-3) days, preferably in the morning. The recommended dose of BMN 190 is according to the participant's age: Birth to < 6 months: 100 mg, 6 months to < 1 year: 150 mg, 1 year to < 2 years: 200 mg (first four doses), 300 mg (subsequent doses) >=2 years: 300 mg. The treatment continued for the duration of at least 144 weeks or until all procedures were completed or the participant discontinued from the study.
  BMN 190 recombinant human tripeptidyl peptidase-1 (rhTPP1)
  Intracerebroventricular access device: Surgical implantation of an MRI compatible ICV access device in the lateral ventricle of the right hemisphere is required for administration of study drug.
- Natural History Comparator: 190-901 Participants: The NH comparator population consisted of subjects from the DEM-CHILD database who satisfied the 190-203 inclusion criteria. The Study 190-901 evaluable population was required to have:
  * At least one assessment ML >= 3
  * At least two ML assessments in the range 1 - 6 and at least 6 months apart
Period: Overall Study
Arm/Group | BMN 190-203 | Natural History Comparator: 190-901 Participants
Started | 14 | 29
Completed | 13 | 29
Not Completed | 1 | 0
Not completed — Participant chose to receive commercial drug in their home country | 1 | 0

BASELINE CHARACTERISTICS:
Population: The 901 subjects weighted according to number of matches: weights for 3, 2, and 1 study 901 subject matched to a given study 203 subject are 1/3,1/2, and 1 times N901/N203 respectively. N901 is the number of 901 subjects matched to 203 subjects (i.e. 29) and N203 is the number of 203 subjects who had matches (i.e. 12). The 203 subjects who had matches were assigned the weight of 1. The common alleles are c.509-1G and c.622C>T
Groups:
- Natural History Comparator:190-901 Participants: The NH comparator population consisted of subjects from the DEM-CHILD database who satisfied the 190-203 inclusion criteria. The Study 190-901 evaluable population was required to have:
  * At least one assessment ML >= 3
  * At least two ML assessments in the range 1 - 6 and at least 6 months apart
- Total: Total of all reporting groups
Arm/Group | BMN 190-203 | Natural History Comparator:190-901 Participants | Total
Number analyzed (Participants) | 12 | 29 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] — The 901 subjects weighted according to number of matches: weights for 3, 2, and 1 study 901 subject matched to a given study 203 subject are 1/3,1/2, and 1 times N901/N203 respectively. N901 is the number of 901 subjects matched to 203 subjects (i.e. 29) and N203 is the number of 203 subjects who had matches (i.e. 12). The 203 subjects who had matches were assigned the weight of 1. The common alleles are c.509-1G and c.622C>T
  years | 2.7 (1.12) | 2.7 (1.09) | 2.7 (1.09)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Percentages were calculated using total no. subjects in ITT Population & in matched subjects as denominators separately
  Number of subjects for Natural history study was rounded to nearest whole no.
  The 901 subjects weighted according to no. of matches: weights for 3, 2,&1 study 901 subject matched to a given study 203 subject are 1/3,1/2, & 1 times N901/N203 respectively. N901 is number of 901 subjects matched to 203 subjects (i.e. 29) & N203 is number of 203 subjects who had matches (i.e. 12). 203 subjects who had matches were assigned weight of 1. Common alleles are c.509-1G & c.622C>T
  Participants
    Female | 8 | 15 | 23
    Male | 4 | 14 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — The 901 subjects weighted according to number of matches: weights for 3, 2, and 1 study 901 subject matched to a given study 203 subject are 1/3,1/2, and 1 times N901/N203 respectively. N901 is the number of 901 subjects matched to 203 subjects (i.e. 29) and N203 is the number of 203 subjects who had matches (i.e. 12). The 203 subjects who had matches were assigned the weight of 1. The common alleles are c.509-1G and c.622C>T
  Participants
    Hispanic or Latino | 1 | 0 | 1
    Not Hispanic or Latino | 11 | 0 | 11
    Unknown or Not Reported | 0 | 29 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — The 901 subjects weighted according to number of matches: weights for 3, 2, and 1 study 901 subject matched to a given study 203 subject are 1/3,1/2, and 1 times N901/N203 respectively. N901 is the number of 901 subjects matched to 203 subjects (i.e. 29) and N203 is the number of 203 subjects who had matches (i.e. 12). The 203 subjects who had matches were assigned the weight of 1. The common alleles are c.509-1G and c.622C>T
  Participants
    White | 12 | 0 | 12
    Unknown or Not Reported | 0 | 29 | 29
CLN2 motor-language (ML) score [Mean (Standard Deviation); unit: score on a scale] — The combined motor/gait and language (ML) score, as derived from the Hamburg CLN2 rating scale, immediately preceding the first infusion. The combined ML score is determined as the sum of the 0-3 point motor (M) and language (L) subscales where 0 represents no function, and 3 represents normal function, and can range from 0 (severely impaired) to 6 (normal). Thus, high scores describe better function & low scores describe poor function
  score on a scale | 5.0 (1.41) | 5.0 (1.38) | 5.0 (1.37)
CLN2 motor scale score at Baseline [Mean (Standard Deviation); unit: score on a scale] — The 901 subjects weighted according to No.of matches:weights for 3,2,&1 study 901 subject matched to a given study 203 subject are 1/3,1/2,&1 times N901/N203 respectively. N901 is No. of 901 subjects matched to 203 subjects(ie 29)& N203 is No.of 203 subjects who had matches(ie12)203 subjects who had matches were assigned weight of 1. Common alleles are c.509-1G & c.622C>T
  The 0-3 point motor(M) subscales, as derived from the Hamburg CLN2 rating scale, where 0 represents no function,& 3 represents normal function.Thus,high scores describe better function & low scores describe poor function
  score on a scale | 2.4 (0.79) | 2.6 (0.54) | 2.6 (0.63)
CLN2 language scale score at Baseline [Mean (Standard Deviation); unit: Score on a scale] — The 901 subjects weighted according to No.of matches:weights for 3,2,&1 study 901 subject matched to a given study 203 subject are 1/3,1/2,&1 times N901/N203 respectively.N901 is No.of 901 subjects matched to 203 subjects(ie 29)& N203 is No.of 203 subjects who had matches(ie12). 203 subjects who had matches were assigned weight of 1. Common alleles are c.509-1G & c.622C>T
  0-3 point language (L) subscales, as derived from the Hamburg CLN2 rating scale, where 0 represents no function, & 3 represents normal function.Thus, high scores describe better function & low scores describe poor function
  Score on a scale | 2.6 (0.67) | 2.4 (0.93) | 2.4 (0.86)
CLN2 motor-language-vision-seizure (MLVS) score [Mean (Standard Deviation); unit: Score on a scale] — The combined motor-language-vision-seizure (MLVS) score as derived from the Hamburg CLN2 rating scale, is determined as the sum of the 0-3 point motor (M) and language (L) vision (V) and seizure (S) subscales where 0 represents no function, and 3 represents normal function, and can range from 0 (severely impaired) to 12 (normal). Thus, high scores describe better function & low scores describe poor function. Population: One subject in the natural history group had missing baseline values for the vision and seizure domains. Therefore MLVS score could not be calculated.
  Score on a scale
    number analyzed (Participants) | 12 | 28 | 40
    (all) | 10.9 (1.56) | 10.2 (2.70) | 10.4 (2.42)
Age at disease onset (years) [Mean (Standard Deviation); unit: years] — The 901 subjects weighted according to number of matches: weights for 3, 2, and 1 study 901 subject matched to a given study 203 subject are 1/3,1/2, and 1 times N901/N203 respectively. N901 is the number of 901 subjects matched to 203 subjects (i.e. 29) and N203 is the number of 203 subjects who had matches (i.e. 12). The 203 subjects who had matches were assigned the weight of 1. The common alleles are c.509-1G and c.622C>T Population: Age at disease onset was missing for several subjects in both 190-203 and the natural history comparator.
  years
    number analyzed (Participants) | 5 | 11 | 16
    (all) | 2.1 (0.82) | 2.6 (0.82) | 2.5 (0.83)

OUTCOME MEASURES:

1. Primary Outcome: Motor Language (ML) Scale: Rate of Decline in the 0 to 6-point ML Score.
Description: Rate of decline in 0 to 6-point ML score, & primary analysis was based on up to 3-1 matching of Study 190-901 evaluable participants with Study 190-203 ITT participants.
  Rate of decline =(-1)x(48x7)x(Ending score - Starting score)/(Ending date - Starting date)
  A positive rate of decline means that subject declined, a negative rate of decline means that subject improved.
  The combined motor/gait and language (ML) score, as derived from Hamburg CLN2 rating scale, immediately preceding first infusion. The combined ML score is determined as sum of 0-3 point motor(M) & language(L) subscales where 0 represents no function, & 3 represents normal function, & can range from 0(severely impaired) to 6(normal). Thus,high scores describe better function & low scores describe poor function.
  The starting assessment is baseline ML assessment & ending assessment is last ML score >0. Note for Study 190-901, baseline ML assessment is defined as assessment of matching to Study 190-203 subj.
Time Frame: Baseline to Last assessment (Week 169)
Population: Matched ITT BMN 190-203: Two subjects in 190-203 ITT population (N=14) were excluded from the 190-203 ITT analysis with matching (N=12) who did not match with any 190-901 subjects on the matching criteria. The matching criteria at baseline were: • Equal ML score • Age within 3 months • Genome: equal number of common alleles (c.622C→T, c.509.1G→C)
  Matched 190-901 Natural history population: 29 subjects from DEM-CHILD database satisfying the criteria listed in the Arm/Group description.
Measure: Mean (Standard Deviation); unit: change in score/48 wk
Arm/Group | BMN 190-203 | Natural History Comparator: 190-901 Participants
Number analyzed (Participants) | 12 | 29
change in score/48 wk | 0.15 (0.243) | 1.30 (0.857)
Statistical Analysis 1: Comparison: BMN 190-203 vs Natural History Comparator: 190-901 Participants; Test type: Superiority — The two-sample T-test with unequal variance was conducted at a significance level of 0.05; p < 0.0001, t-test, unequal variance

2. Primary Outcome: Probability of Unreversed 2-Point Decline in Motor-language (ML) Score or Score of 0
Description: An unreversed 2-point decline is any decline of 2 points or more that had not reversed to a 1-point decline (or better) at last recorded observation. An unreversed score of 0 is a decline to 0 that had not increased to a score >0 at last recorded observation
  ML score decline is measured by motor & language domains on CLN2 rating scale. Combined motor/gait &language (ML) score, as derived from Hamburg CLN2 rating scale, immediately preceding first infusion. Combined ML score is determined as sum of the 0-3 point motor(M)&language(L) where 0 represents no function, & 3 represents normal function, & can range from 0 (severely impaired) to 6 (normal). Thus, high scores describe better function & low scores describe poor function
  Model includes data up to week 169. Estimates from the model are presented for Wks 49, 97 & 145
  No.analyzed is no.of subj out of overall no.of participants analyzed who have not been censored/had unreversed 2-point decline/score of 0 at given time points.
Time Frame: Baseline to Last assessment (Week 169)
Population: Matched ITT BMN 190-203: Two subjects in 190-203 ITT Population(N=14) were excluded from the 190-203 ITT analysis with matching (N=12) who did not match with any 190-901 subjects on the matching criteria. The matching criteria at baseline were: Equal ML score, age within 3 months and genome with equal number of common alleles(c.622C→T, c.509.1G→C).
  Matched 190-901 Natural history population: 29 subjects from DEM-CHILD database satisfying the criteria listed in the Arm/Group description.
Measure: Number (95% Confidence Interval); unit: Probability of decline
Arm/Group | BMN 190-203 | Natural History Comparator: 190-901 Participants
Number analyzed (Participants) | 12 | 29
Probability of decline
  Probability of decline: Week 49: number analyzed (Participants) | 12 | 23
  Probability of decline: Week 49 | 0.0 [0.00 to 0.00] | 0.141 [0.05 to 0.35]
  Probability of decline: Week 97: number analyzed (Participants) | 11 | 16
  Probability of decline: Week 97 | 0.083 [0.01 to 0.46] | 0.397 [0.23 to 0.62]
  Probability of decline: Week 145: number analyzed (Participants) | 10 | 6
  Probability of decline: Week 145 | 0.167 [0.04 to 0.52] | 0.774 [0.59 to 0.92]
Statistical Analysis 1: Comparison: BMN 190-203 vs Natural History Comparator: 190-901 Participants; Test type: Superiority; p < .0001, Cox Model Wald Test; Hazard Ratio (HR) = 0.091, 95% CI 2-sided [0.021 to 0.393] — Hazard ratio is based on Cox proportional hazards model with a factor of study group

3. Primary Outcome: Probability of Decline of Unreversed Motor-language (ML) Score of 0
Description: The combined motor/gait and language (ML) score, as derived from the Hamburg CLN2 rating scale, immediately preceding the first infusion. The combined ML score is determined as the sum of the 0-3 point motor (M) and language (L) subscales where 0 represents no function, and 3 represents normal function, and can range from 0 (severely impaired) to 6 (normal). Thus, high scores describe better function and low scores describe poor function.
  Model includes data up to week 169. Estimates from the model are presented for Weeks 49, 97 and 145.
  No.analyzed is no.of subj out of overall no.of participants analyzed who have not been censored/had unreversed decline/score of 0 at given time points
Time Frame: Baseline to Last assessment (Week 169)
Population: Matched ITT BMN 190-203: Two subjects in 190-203 ITT Population (N=14) were excluded from the 190-203 ITT analysis with matching (N=12) who did not match with any 190-901 subjects on the matching criteria. The matching criteria at baseline were: Equal ML score, age within 3 months and genome with equal number of common alleles (c.622C→T, c.509.1G→C).
  Matched 190-901 Natural history population: 29 subjects from DEM-CHILD database satisfying the criteria listed in the Arm/Group description
Measure: Number (95% Confidence Interval); unit: Probability of decline
Arm/Group | BMN 190-203 | Natural History Comparator: 190-901 Participants
Number analyzed (Participants) | 12 | 29
Probability of decline
  Probability of decline: Week 49: number analyzed (Participants) | 12 | 26
  Probability of decline: Week 49 | 0.0 [0.00 to 0.00] | 0.03 [0.00 to 0.26]
  Probability of decline: Week 97: number analyzed (Participants) | 12 | 22
  Probability of decline: Week 97 | 0.0 [0.00 to 0.00] | 0.149 [0.06 to 0.37]
  Probability of decline: Week 145: number analyzed (Participants) | 12 | 13
  Probability of decline: Week 145 | 0.0 [0.00 to 0.00] | 0.336 [0.18 to 0.57]
Statistical Analysis 1: Comparison: BMN 190-203 vs Natural History Comparator: 190-901 Participants; Test type: Superiority; p = 0.0032, Cox Model Wald Test; Hazard Ratio (HR) = 0.000, 95% CI 2-sided [0.000 to 0.000] — Hazard ratio is based on Cox proportional hazards model with a factor of study group

4. Primary Outcome: Rate of Decline in Individual Motor Domains
Description: Rate of decline = (-1) x (48 x 7) x (Ending score - Starting score)/(Ending date - Starting date).
  A positive rate of decline means that the subject declined, a negative rate of decline means that the subject improved.
  The 0-3 point motor (M) subscales, as derived from the Hamburg CLN2 rating scale, where 0 represents no function, and 3 represents normal function. Thus, high scores describe better function, and low scores describe poor function.
Time Frame: Baseline to Last assessment (Week 169)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: change in score/48 wk
Arm/Group | BMN 190-203 | Natural History Comparator: 190-901 Participants
Number analyzed (Participants) | 12 | 29
change in score/48 wk | 0.05 (0.120) | 0.59 (0.496)
Statistical Analysis 1: Comparison: BMN 190-203 vs Natural History Comparator: 190-901 Participants; Test type: Superiority; p < .0001, t-test, unequal variance

5. Primary Outcome: Rate of Decline in Individual Language Domains
Description: Rate of decline = (-1) x (48 x 7) x (Ending score - Starting score)/(Ending date - Starting date).
  A positive rate of decline means that the subject declined, a negative rate of decline means that the subject improved.
  The 0-3 point language (L) subscales, as derived from the Hamburg CLN2 rating scale, where 0 represents no function, and 3 represents normal function. Thus, high scores describe better function and low scores describe poor function.
  Patients with baseline score of 0 are excluded.
Time Frame: Baseline to Last assessment (Week 169)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: change in score/48 wk
Arm/Group | BMN 190-203 | Natural History Comparator: 190-901 Participants
Number analyzed (Participants) | 12 | 28
change in score/48 wk | 0.10 (0.146) | 0.77 (0.715)
Statistical Analysis 1: Comparison: BMN 190-203 vs Natural History Comparator: 190-901 Participants; Test type: Superiority; p < .0001, t-test, unequal variance

6. Secondary Outcome: Probability of Decline of Disease Manifestation at Week 49 & 97
Description: Disease manifestation is defined as post-baseline consecutive measurements of M,L,V/S scores<3, measured atleast 22days apart.
  Combined motor-language-vision-seizure(MLVS)score as derived from Hamburg CLN2 rating scale, is determined as sum of 0-3 point motor(M)language(L)visio(V)&seizure(S) subscales where 0 represents no function,&3 represents normal function,&can range from 0(severely impaired)to12(normal).Thus, high scores describe better function & low scores describe poor function.
  901 subj weighted according to no.of matches:weights for 3,2,&1 study 901 subj matched to a given study 203 subj are 1/3,1/2, &1 times N901/N203 respectively. N901 is no.of 901 subj matched to 203 subj(ie.18)&N203 is no.203 subj who had matches (i.e.7).203 subj who had matches were assigned weight of 1.
  No.analyzed is no.of subj out of overall no.of participants analyzed who have not been censored/had decline of disease manifestation at given time points
Time Frame: Baseline to Last assessment (Week 169)
Population: Matched ITT BMN190-203:2 subj in190-203 ITT Population(N=14)were excluded from 190-203 ITT analysis with matching(N=12)who did not match with any190-901 subj on matching criteria.Matching criteria at baseline were:Equal ML score,age<3 months&genome with equal no.of common alleles(c.622C→T,c.509.1G→C).
  Matched190-901 Natural history population:29 subj from DEM-CHILD database satisfying criteria listed in Arm descp
  Model includes data upto wk169.Estimates from model are presented for Wks 49&97
Measure: Number (95% Confidence Interval); unit: Probability of decline
Arm/Group | BMN 190-203 | Natural History Comparator: 190-901 Participants
Number analyzed (Participants) | 7 | 18
Probability of decline
  Probability of decline: Week 49: number analyzed (Participants) | 6 | 11
  Probability of decline: Week 49 | 0.143 [0.02 to 0.67] | 0.405 [0.22 to 0.67]
  Probability of decline: Week 97: number analyzed (Participants) | 5 | 4
  Probability of decline: Week 97 | 0.286 [0.08 to 0.74] | 0.762 [0.55 to 0.93]
Statistical Analysis 1: Comparison: BMN 190-203 vs Natural History Comparator: 190-901 Participants; Test type: Superiority; p = 0.0081, Cox Model Wald Test; The p value is a test that the hazard ratio equal to 1; Hazard Ratio (HR) = 0.209, 95% CI 2-sided [0.059 to 0.735] — Hazard ratio is based on Cox proportional hazards model with a factor of study group. Hazard Ratio (HR) 190-203 vs DEM-CHILD

7. Secondary Outcome: Probability of Decline of Disease Manifestation at Week 145
Description: Disease manifestation is defined as post-baseline consecutive measurements of M,L,V/S scores<3,measured atleast 22days apart
  Combined MLVS score,as derived from Hamburg CLN2 rating scale,is determined as sum of 0-3 point motor(M)language(L)vision(V)&seizure(S) subscales where 0 represents no function,&3 represents normal function,&can range from 0(severely impaired) to 12(normal).Thus,high scores describe better function&low scores describe poor function
  901 subj weighted according to no.of matches:weights for 3,2,&1 study 901 subj matched to given study 203 subj are 1/3,1/2, &1 times N901/N203 respectively.N901 is no.of 901 subj matched to 203 subj(ie.18)&N203 is no.203 subj who had matches(i.e.7).203 subj who had matches were assigned weight of 1
  Model includes data upto wk169.Estimates from model are presented for Wk145
  No.analyzed is no.of subj out of overall no.of participants analyzed who have not been censored/had decline of disease manifestation at given time point
Time Frame: Baseline to Week 145
Population: Matched ITT BMN190-203:2 subj in 190-203 ITT Pop(N=14) were excluded from 190-203 ITT analysis with matching(N=12) who did not match with any 190-901 subj on matching criteria. Matching criteria at baseline were:Equal ML score, age within 3 months & genome with equal no. of common alleles(c.622C→T, c.509.1G→C).
  Matched 190-901 Natural history pop:29 subj from DEM-CHILD database satisfying criteria listed in Arm/Group descp.
  No.of subj analyzed for 190-901=0 & hence this arm is not included
Measure: Number (95% Confidence Interval); unit: Probability of decline
Arm/Group | BMN 190-203
Number analyzed (Participants) | 4
Probability of decline | 0.429 [0.16 to 0.83]

8. Secondary Outcome: Change From Baseline in ML Scale Score
Description: The combined motor/gait and language (ML) score, as derived from the Hamburg CLN2 rating scale, immediately preceding the first infusion. The combined ML score is determined as the sum of the 0-3 point motor (M) and language (L) subscales where 0 represents no function, and 3 represents normal function, and can range from 0 (severely impaired) to 6 (normal). Thus, high scores describe better function and low scores describe poor function.
  Some participants did not have follow-up at all time points.
Time Frame: Baseline to Week 49, Week 97, Week 145, & Week 169
Population: 190-901 participants weighted according to no. of matches: weights for 3,2,&1 study 190-901 participant matched to a given Study190-203 participant were1/3,1/2,&1 times N901/N203, respectively. N901 was no. of 190-901 participants matched to 190-203 participants (ie,29) &N203 was no. of 190-203 participants who had matches (ie,12).190-203 participants who had matches were assigned weight of 1.
  Each participant in Study 190-901 had their scores imputed to time points using linear interpolation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BMN 190-203 | Natural History Comparator: 190-901 Participants
Number analyzed (Participants) | 12 | 29
score on a scale
  Change from Baseline to Week 49: number analyzed (Participants) | 12 | 27
  Change from Baseline to Week 49 | -0.0 (0.57) | -0.8 (1.05)
  Change from Baseline to Week 97: number analyzed (Participants) | 12 | 25
  Change from Baseline to Week 97 | 0.0 (0.43) | -1.6 (1.22)
  Change from Baseline to Week 145: number analyzed (Participants) | 12 | 21
  Change from Baseline to Week 145 | -0.4 (0.78) | -3.1 (1.61)
  Change from Baseline to Week 169: number analyzed (Participants) | 11 | 9
  Change from Baseline to Week 169 | -0.4 (0.67) | -3.7 (2.39)

9. Secondary Outcome: Changes From Baseline in MLV Scale Score
Description: The combined motor-language-vision (MLV) score, as derived from the Hamburg CLN2 rating scale, is determined as the sum of the 0-3 point motor (M), language (L) & vision (V) subscales where 0 represents no function, and 3 represents normal function, and can range from 0 (severely impaired) to 9 (normal). Thus, high scores describe better function and low scores describe poor function.
  Some participants did not have follow-up at all time points.
Time Frame: Baseline to Week 49, Week 97, Week 145, & Week 169
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BMN 190-203 | Natural History Comparator: 190-901 Participants
Number analyzed (Participants) | 12 | 29
score on a scale
  Change from Baseline to Week 49: number analyzed (Participants) | 12 | 27
  Change from Baseline to Week 49 | -0.1 (0.74) | -1.0 (1.31)
  Change from Baseline to Week 97: number analyzed (Participants) | 12 | 25
  Change from Baseline to Week 97 | -0.1 (0.51) | -2.1 (1.71)
  Change from Baseline to Week 145: number analyzed (Participants) | 12 | 21
  Change from Baseline to Week 145 | -0.7 (1.06) | -3.9 (1.98)
  Change from Baseline to Week 169: number analyzed (Participants) | 11 | 9
  Change from Baseline to Week 169 | -0.7 (1.10) | -4.5 (3.04)

10. Secondary Outcome: Changes From Baseline in the 0-12 Point MLVS Motor, Language, Vision, and Seizure Subscales (MLVS) Score.
Description: The combined motor-language-vision-seizure (MLVS) score, as derived from the Hamburg CLN2 rating scale, is determined as the sum of the 0-3 point motor (M) and language (L) vision (V) and seizure (S) subscales where 0 represents no function, and 3 represents normal function, and can range from 0 (severely impaired) to 12 (normal). Thus, high scores describe better function and low scores describe poor function.
  Some participants did not have follow-up at all time points.
Time Frame: Baseline to Week 49, Week 97, Week 145, & Week 169
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BMN 190-203 | Natural History Comparator: 190-901 Participants
Number analyzed (Participants) | 12 | 29
score on a scale
  Change from Baseline to Week 49: number analyzed (Participants) | 12 | 26
  Change from Baseline to Week 49 | -0.2 (0.86) | -1.5 (1.39)
  Change from Baseline to Week 97: number analyzed (Participants) | 12 | 24
  Change from Baseline to Week 97 | -0.1 (0.51) | -3.0 (1.78)
  Change from Baseline to Week 145: number analyzed (Participants) | 12 | 21
  Change from Baseline to Week 145 | -0.6 (0.99) | -5.5 (2.48)
  Change from Baseline to Week 169: number analyzed (Participants) | 11 | 9
  Change from Baseline to Week 169 | -0.6 (1.03) | -6.4 (3.43)

11. Secondary Outcome: Percentage Change From Baseline to Last Assessment: Volume of Cerebrospinal Fluid (mL)
Time Frame: Baseline to Last assessment (Week 169)
Population: Intent-to-treat (ITT) population.
  One subject did not have any follow-up MRI data available.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | BMN 190-203
Number analyzed (Participants) | 13
Percentage | 0.7 (13.18)

12. Secondary Outcome: Percentage Change From Baseline to Last Assessment: Volume of Total Cortical Gray Matter (mL)
Time Frame: Baseline to Last assessment (Week 169)
Population: Intent-to-treat (ITT) population.
  One subject did not have any follow-up MRI data available.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | BMN 190-203
Number analyzed (Participants) | 13
Percentage | -10.3 (13.86)

13. Secondary Outcome: Percentage Change From Baseline to Last Assessment: Volume of Total White Matter (mL)
Time Frame: Baseline to Last assessment (Week 169)
Population: Intent-to-treat (ITT) population.
  One subject did not have any follow-up MRI data available.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | BMN 190-203
Number analyzed (Participants) | 13
Percentage | 5.4 (20.86)

14. Secondary Outcome: Change From Baseline to Last Assessment: Whole Brain Apparent Diffusion Coefficient Value
Description: The apparent diffusion coefficient (ADC) represents the calculated diffusion coefficient of water molecules in the direction of the applied gradients measured during diffusion MRI, a technique used to explore the architecture and microstructural properties of both the white and gray matter of the brain.
Time Frame: Baseline to Last assessment (Week 169)
Population: Intent-to-treat (ITT) population.
  One subject did not have any follow-up MRI data available.
Measure: Mean (Standard Deviation); unit: mm^2/s
Arm/Group | BMN 190-203
Number analyzed (Participants) | 13
mm^2/s | 0.0 (0.04)

ADVERSE EVENTS:
Time Frame: Up-to Safety Follow-Up (6 months after last dose).
Description: Atrioventricular block 2nddegree was assessed non-serious by inv but was later upgraded to serious by BioMarin.Inv assessed event as not related to BMN190;however,due to absence of alternative etiological factors&strong temporal relationship,BioMarin conservatively assessed event possibly related to BMN190.This event was considered a suspected unexpected serious adverse reaction(SUSAR)
  AEs&death were collected for BMN190-203 study but it was not collected for BMN190-901(Natural History study)
Groups:
- BMN 190 Recombinant Human Tripeptidyl Peptidase-1 (rhTPP1): BMN 190 was administered by continuous Intracerebroventricular (ICV) infusion at the rate of 2.5 mL/hour for approximately 4 hours every 14 (+/-3) days, preferably in the morning. The recommended dose of BMN 190 is according to the participant's age: Birth to < 6 months: 100 mg, 6 months to < 1 year: 150 mg, 1 year to < 2 years: 200 mg (first four doses), 300 mg (subsequent doses) >=2 years: 300 mg. The treatment continued for the duration of at least 144 weeks or until all procedures were completed or the participant discontinued from the study.
  BMN 190 recombinant human tripeptidyl peptidase-1 (rhTPP1)
  Intracerebroventricular access device: Surgical implantation of an MRI compatible ICV access device in the lateral ventricle of the right hemisphere is required for administration of study drug.
Arm/Group | BMN 190 Recombinant Human Tripeptidyl Peptidase-1 (rhTPP1)
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 12/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 190 Recombinant Human Tripeptidyl Peptidase-1 (rhTPP1) (N=14)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1)
Pyrexia (General disorders) | 4 (7)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Mycoplasma infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (3)
Pyelonephritis (Infections and infestations) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (2)
Gastrointestinal fistula (Gastrointestinal disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Complication of device insertion (General disorders) | 1 (1)
Medical device site haematoma (General disorders) | 1 (1)
Medical device site irritation (General disorders) | 1 (1)
Influenza (Infections and infestations) | 2 (3)
Corona virus infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Pleocytosis (Nervous system disorders) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1)
Propionibacterium test positive (Investigations) | 1 (1)
Device leakage (Product Issues) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN 190 Recombinant Human Tripeptidyl Peptidase-1 (rhTPP1) (N=14)
Pyrexia (General disorders) | 12 (62)
Upper respiratory tract infection (Infections and infestations) | 12 (26)
Extensor plantar response (Nervous system disorders) | 7 (7)
Gastroenteritis (Infections and infestations) | 7 (10)
Generalised tonic-clonic seizure (Nervous system disorders) | 6 (18)
Vomiting (Gastrointestinal disorders) | 5 (7)
Contusion (Injury, poisoning and procedural complications) | 4 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (9)
Dysphagia (Gastrointestinal disorders) | 4 (5)
Hypersensitivity (Immune system disorders) | 4 (20)
Influenza (Infections and infestations) | 4 (6)
Medication monitoring error (Injury, poisoning and procedural complications) | 4 (4)
Atonic seizures (Nervous system disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 3 (3)
Corona virus infection (Infections and infestations) | 3 (4)
Device leakage (Product Issues) | 3 (4)
Dystonia (Nervous system disorders) | 3 (3)
Partial seizures (Nervous system disorders) | 3 (28)
Rash (Skin and subcutaneous tissue disorders) | 3 (4)
Rhinitis (Infections and infestations) | 3 (5)
Seizure (Nervous system disorders) | 3 (8)
Speech disorder developmental (Nervous system disorders) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bronchitis (Infections and infestations) | 2 (3)
Dental caries (Gastrointestinal disorders) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (5)
Dyskinesia (Nervous system disorders) | 2 (34)
Epilepsy (Nervous system disorders) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (8)
Foreign body (Injury, poisoning and procedural complications) | 2 (3)
Insomnia (Psychiatric disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Needle issue (Product Issues) | 2 (3)
Otitis media (Infections and infestations) | 2 (2)
Parainfluenzae virus infection (Infections and infestations) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (3)
Sleep disorder (Psychiatric disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Tonsillitis (Infections and infestations) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Viral test positive (Investigations) | 2 (2)
Visual impairment (Eye disorders) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Athetosis (Nervous system disorders) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 (1)
Bicuspid aortic valve (Congenital, familial and genetic disorders) | 1 (1)
Body temperature increased (Investigations) | 1 (4)
CSF red blood cell count positive (Investigations) | 1 (1)
Chills (General disorders) | 1 (1)
Complication of device insertion (General disorders) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1)
Device breakage (Product Issues) | 1 (1)
Device malfunction (Product Issues) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Ear haemorrhage (Ear and labyrinth disorders) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Electrocardiogram abnormal (Investigations) | 1 (1)
Electroencephalogram abnormal (Investigations) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (2)
Exanthema subitum (Infections and infestations) | 1 (1)
Eye movement disorder (Eye disorders) | 1 (11)
Eyelid contusion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Febrile convulsion (Nervous system disorders) | 1 (2)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1)
Gait disturbance (General disorders) | 1 (2)
Gastrointestinal fistula (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Hepatic enzyme increased (Investigations) | 1 (2)
Hordeolum (Infections and infestations) | 1 (3)
Human rhinovirus test positive (Investigations) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Language disorder (Nervous system disorders) | 1 (2)
Laryngitis (Infections and infestations) | 1 (1)
Malaise (General disorders) | 1 (1)
Medical device site haematoma (General disorders) | 1 (1)
Medical device site irritation (General disorders) | 1 (1)
Medical device site swelling (General disorders) | 1 (1)
Mycoplasma infection (Infections and infestations) | 1 (1)
Myoclonic epilepsy (Nervous system disorders) | 1 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Pain (General disorders) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Partial seizures with secondary generalisation (Nervous system disorders) | 1 (2)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (2)
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Petit mal epilepsy (Nervous system disorders) | 1 (3)
Pharyngitis (Infections and infestations) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1)
Pleocytosis (Nervous system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (3)
Pneumonia chlamydial (Infections and infestations) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Propionibacterium test positive (Investigations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Pyuria (Infections and infestations) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1)
Respiratory syncytial virus test (Investigations) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (2)
Respirovirus test positive (Investigations) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1)
Rotavirus infection (Infections and infestations) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)
Seizure cluster (Nervous system disorders) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Talipes (Congenital, familial and genetic disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restrictions on the PI are that (i) they cannot publish results communications until after the multicenter dataset is published, (ii) the sponsor has an opportunity to review results communications prior to public release, and (iii) the sponsor can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days.

DOCUMENTS (2):
  • Study Protocol (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/89/NCT02678689/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/89/NCT02678689/SAP_001.pdf